CLINICAL TRIAL: NCT05224310
Title: Comparing the Quality of Analgesia With Ultrasound-guided Pectoral Nerve Block and Serratus Plane Block in Patients Undergoing Modified Radical Mastectomy
Brief Title: Comparing the Quality of Analgesia With Pectoral Nerve Block and Serratus Plane Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PECS vs SAP
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Mastectomy; Breast Cancer
Keywords: analgesia; postoperative pain; PECS block; SAP block
MeSH Terms: conditions — Breast Neoplasms; Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectoral nerve block (Active Comparator): Starting from the lateral third of the clavicle and moving distally and laterally to the midaxillary line. The pectoral major and minor muscles will be identified and 10 mL of bupivacaine 0.25% will be injected between the 2 muscles, and then move the ultrasound probe towards the axilla until the serratus anterior is identified above the second, third, and fourth ribs then injection of 20 mL of bupivacaine 0.25% after negative aspiration into the fascial plane between pectoralis minor and serratus anterior muscles.
  Interventions: Procedure: PECS block, SAP block
- Serratus anterior plane block (Active Comparator): Aiming to find the serratus anterior muscle the investigator will identify the fifth rib in the midaxillary line by the linear probe in the sagittal plane. The latissimus dorsi muscle (superficial and posterior), teres major muscle (superior) and serratus muscles (deep and inferior) will be detected using ultrasound.
  The investigator will penetrate the serratus anterior muscle by a 23 GA, 35 mm needle in-plane to ultrasound probe from supero-anterior to postero-inferior to inject deep to it.
  Interventions: Procedure: PECS block, SAP block

INTERVENTIONS:
Procedure: PECS block, SAP block — performing either PECS block or SAP block

SUMMARY:
The use of pectoral nerve block (PECSB) is a new technique during modified radical mastectomy MRM.

The Serratus anterior Plane (SAP) Block has been proven to be an effective component of multimodal analgesia regimens for a variety of thoracic procedures including MRM.

In this study, the investigators will assess and compare the quality of analgesia with ultrasound-guided Serratus plane block and pectoral nerve block in patients undergoing modified radical mastectomy MRM.

DETAILED DESCRIPTION:
Breast cancer is the most common cause of cancer death among women worldwide. In Egypt, breast cancer is the most common malignancy in women, accounting for 38.8% of cancers in this population. It is estimated that the breast cancer mortality rate is around 11%, being the second cause of cancer-related mortality after liver cancer.

According to the European network of cancer registries, most breast cancer patients require breast surgery to remove the primary tumour and axillary staging or dissection. Approximately 40% of these patients will experience clinically significant acute postoperative pain. Furthermore, acute postoperative pain is an important risk factor for the development of persistent chronic postoperative pain in women after breast surgery.

Acute postoperative pain is associated with increased comorbidity and hospital stay length; as it will affect respiratory functions, chest wall compliance, cardiac output, blood pressure, cardiac workload, metabolism, oxygen consumption, decreased tone of gastrointestinal and urinary tracts and marked increases in catabolic hormones (catecholamine, adrenocorticotrophic hormone, antidiuretic hormone, glucagon, and aldosterone) while decreasing anabolic hormones such as insulin and testosterone.

It has been reported that up to half of the patients have a negative impact of pain on their activities and up to one-quarter report moderate to high impact on their daily activities at home and work. Thus, more effective treatment modalities are used for decreasing postoperative pain in mastectomy patients include; patient-controlled analgesia PCA, thoracic epidural, and thoracic paravertebral block.

While the key requirement for successful regional anaesthetic blocks is ensuring optimal distribution of local anaesthetic around nerve structures, ultrasound guidance enables the anaesthetist to secure an accurate needle position and to monitor the distribution of the local anaesthetic in real-time.

It was found that blockade of the lateral cutaneous branches of thoracic intercostal nerves (T2-T12) will provide analgesia to the anterolateral chest wall in most patients.

The Serratus anterior Plane (SAP) Block has proven to be an effective component of multimodal analgesia regimens for a variety of thoracic procedures. It is designed to block primarily the thoracic intercostal nerves and to provide complete analgesia of the lateral part of the thorax and it may be a viable alternative to paravertebral blockade and thoracic epidural analgesia and may be associated with fewer side effects. It's straightforward to perform, with a high success rate and minimal incidence of complications. It was reported prolonged numbness over the area supplied by the lateral cutaneous branches of the T2-T9 spinal nerves using only 0.4 ml.kg-1 0.125% levobupivacaine. This is remarkable because alternative techniques such as intercostal, intrapleural and thoracic paravertebral block require relatively high concentrations and volumes of local anaesthetics to produce similarly prolonged, multi-dermatomal thoracic analgesia.

Blanco et al. reported the use of pectoral nerve block (PECSB) as a new technique during modified radical mastectomy MRM. PECSB is an interfascial plane block where local anaesthetics deposited into the plane between the pectoralis major muscle and the pectoralis minor muscle (PECS-I block) and above the serratus anterior muscle at the third rib (PECS-II block) blocking the pectoral, intercostobrachial, intercostals III, IV, V, and VI; and long thoracic nerves. The PECSB is expected to provide analgesia for breast cancer surgery BCS.

In this study, the investigators will assess and compare the quality of analgesia with ultrasound-guided Serratus plane block and pectoral nerve block in patients undergoing modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult, female patients,
* ASA physical status I, II, and III
* Aged older than 18 years
* Scheduled for modified radical mastectomy surgery under general anaesthesia.

Exclusion Criteria:

* Any known allergies to the study drugs.
* Apparent anatomical abnormalities or infections in the serratus region.
* Bleeding disorders e.g. thrombocytopenia, high INR, high PT in the chronic liver or impaired kidney).
* Patients on chronic pain medications or regularly receiving analgesics.
* Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients with breast cancer undergoing modified radical mastectomy surgery under general anaesthesia
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The first request for analgesia | immediately at the end of 24 hours post operatively
  the time from the completion of the block to the time of the first request for analgesia.

SECONDARY OUTCOMES:
Post-operative pain | immediately postoperatively 0,2,4,6,8,12,14,16,18,20,22,and 24 h after surgery at rest
  pain will be evaluated using the "Visual Analogue Scale" at rest, the minimal score is 0 which means no pain at all, and the maximum is 10 which means unbearable pain, a higher score is worse and means a higher perception of pain, and more need for analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Alshawadfy, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt